CLINICAL TRIAL: NCT03057509
Title: A Pilot Study Of Ga-68-DOTA-TOC Imaging In Participants With Small Bowel Carcinoid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Umar Mahmood, Professor of Radiology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-193
Record Dates: First submitted 2017-02-03; First posted 2017-02-20 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Small Bowel Carcinoid Tumor
Keywords: Carcinoid Tumors
MeSH Terms: conditions — Carcinoid Tumor | interventions — gallium Ga 68 dotatate; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Gallium PET/MR Imaging (Experimental): Siemens PET/MR scanner at Martinos Center for Biomedical Imaging will be use.
  * Standard Siemens software will be used to perform image analysis and measure parameters such as SUVmean, SUVmax and MTV.
  * Standard LAR Octreotide will be administered.
  * Ga-68-DOTA-TOC that will be administered prior to PET/MR imaging at 7 days after standard LAR octreotide administration and again at 28 day.
  * Ga-68-DOTA-TOC will be administered as a single intravenous dose at a pre-determine dosage.
  Interventions: Drug: Ga-68-DOTA-TOC; Device: Siemens PET/MR scanner; Other: Standard Siemens Software; Drug: LAR Octreotide

INTERVENTIONS:
Drug: Ga-68-DOTA-TOC — Ga-68-DOTA-TOC is a imaging radiotracer that is used for positron emission tomography imaging of a variety of the neuroendocrine tumors. This radiotracer in the body binds to several subtypes of the somatostatin receptor and accumulates in the tissue with high expression of these receptors. Therefore neuroendocrine tumors that express somatostatin receptors can be imaged using this radiotracer.
Device: Siemens PET/MR scanner — Positron emission tomography-magnetic resonance (PET/MR) is a hybrid imaging technology that incorporates magnetic resonance imaging (MRI) soft tissue morphological imaging and positron emission tomography (PET) functional imaging. The Siemens PET/MR system (Biograph mMR) received a CE mark and FDA approval for clinical diagnostic imaging.
Other: Standard Siemens Software — The Siemens PET/MR scanner are equipped with a standard clinical visualization software with the advanced application tools based on the Siemens image interpretation engine called syngo.via. This software allows for visualization and interpretation of the image data-sets in the clinical environment.
Drug: LAR Octreotide — LAR octreotide is a man-made protein that is similar to a hormone in the body called somatostatin. LAR Octreotide lowers many substances in the body such as insulin and glucagon, growth hormone, and chemicals that affect digestion. LAR octreotide is used to treat a variety of clinical conditions but most importantly to reduce flushing episodes and watery diarrhea caused by cancerous tumors such as neuroendocrine tumors.
  Other Names: Sandostatin

SUMMARY:
This research study is designed to evaluate a type of scan called Ga-68-DOTA-TOC positron emission tomography (PET) scanning as a way of assessing carcinoid tumors.

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study intervention.

Many patients who are diagnosed with carcinoid tumor undergo treatment with long acting release (LAR) octreotide. It is presently standard for all patients to receive equal doses of octreotide. However, the response to the treatment with the same dose of medication may vary substantially from one person to another. This study uses a novel form of PET/MR imaging to try and better understand how to treat carcinoid tumors, and may in the future allow doctors to tailor treatment dosing based on PET/MR findings and select the right drug dose for an individual person. It is important to note that the participant method of treatment and the dose of the participant medication (Octreotide LAR) will not change in this study.

The imaging technique used in this study is called Ga-68-DOTA-TOC PET/MR scanning. Ga-68-DOTA-TOC is a radioactive tracer that is given by vein to participants before PET scanning. The scanner then detects radioactivity from the tracer that is attached to cells within the body and uses this information to create images (pictures) on a computer screen that can then be analyzed.

These types of scans are investigational. "Investigational", meaning that the scans are still being studied and that research doctors are trying to find out more about them. It also means that the FDA (U.S. Food and Drug Administration) has not approved these types of PET scans for this type of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Have histologically or cytologically confirmed small bowel carcinoid tumor
* Receiving a stable dose of octreotide LAR as a part of a treatment regimen for ≥3months
* Presently planned for ongoing octreotide according to current standard of care for at least 18 months (i.e. throughout the study follow-up period).
* Presently planned for restaging using contrast-enhanced CT scans at baseline and at least every 6 months, as a part of their standard of care assessments.
* The effects of Ga-68-DOTA-TOC on the developing human fetus are unknown. For this reason and because PET imaging agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Ga-68-DOTA-TOC administration.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have had radiotherapy within 4 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
* Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions to IV contrasts or reactions attributed to compounds of similar chemical or biologic composition to Ga-68-DOTA-TOC used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because Ga-68-DOTA-TOC have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to administration of Ga-68-DOTA-TOC to mothers, breastfeeding mothers are also excluded from this study.
* Expected lifespan less than 18 months by investigator assessment
* Previous hypersensitivity reaction to LAR octreotide
* Non-removable non-MR compatible placements including hearing aid or dentures, metal IUD, surgical aneurysm clips, cardiac pacemaker, prosthetic heart valve, neurostimulator, implanted pumps, cochlear implants, metal rods, plates or screws, surgery leaving implanted materials, metal injury to eye, metallic tattoos anywhere on the body, tattoos near the eye and transdermal patches
* History of Meniere's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-10-31 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean Change in SUVmax | 2 years
  The mean change of SUVmax from 68Ga-DOTATOC PET scan obtained at peak and trough octreotide LAR therapy.
Mean Change in Total Molecular Burden of The Lesions | 2 Years
  The mean change of Total Molecular Tumor Burden is measured from 68Ga-DOTATOC PET scan obtained at peak and trough octreotide LAR therapy.

SECONDARY OUTCOMES:
Correlation Of Change In Receptor Occupancy With The PFS of patients | 2 years
Progression Free Survival Rate | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Umar Mahmood, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts general Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No